CLINICAL TRIAL: NCT02413918
Title: Open Label Study of Iloperidone (IL) as Adjunctive Treatment in Mixed States (MS) of Bipolar Disorder (BD)
Brief Title: Iloperidone in Mixed States of Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20120137
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2017-05

CONDITIONS: Bipolar Disorder
Keywords: mixed episode
MeSH Terms: conditions — Bipolar Disorder | interventions — iloperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label iloperidone (Experimental): open label iloperidone (oral tablet, 6mg-24mg, QD, 20 weeks) as adjunct to current lithium, divalproex, or lamotrigine.
  Interventions: Drug: iloperidone

INTERVENTIONS:
Drug: iloperidone — Qualifying subjects will take iloperidone starting at 2mg and up to a minimum of 12mg, maximum of 24mg, for 20 weeks in conjunction to the subjects current lithium, and or divalproex, and or lamotrigine.
  Other Names: Fanapt

SUMMARY:
1. To assess the acute and long-term bimodal efficacy of iloperidone (IL), as an adjunct to ongoing treatment with lithium (Li) or divalproex (DIV) or lamotrigine (LAM) or any combination of the three thereof, in a group of patients with an index episode of a mixed state in BD.
2. To assess background, baseline features, and behavioral components which characterize treatment response/non-response in the acute and long term management of MS

DETAILED DESCRIPTION:
This is a prospective 20-week, open-label study of iloperidone added to ongoing treatment regimen with mood stabilizers (Li or DIV or LAM or any combination of these) in the acute and maintenance treatment of MS- Total number of subjects: 40.

Severity of the illness and psychopathological features will be measured by the following rating scales: YMRS, MADRS, CGI-S and GAS, and the BISS .

The study will monitor the safety and tolerability of the combination iloperidone plus mood stabilizers.

Efficacy Measures: Primary efficacy measures include 1) Mixed effects repeat measure of change from baseline in BISS total score and, secondarily, manic and depression subscale scores.

Secondary Efficacy Measures: 1) response defined as 50% reduction in YMRS and MADRS and 2) Time to intervention or discontinuation for any mood episode.

Iloperidone will be initiated at 2 mg at hs on day 1 with increase to 4mg at hs on day 2, 8 mg at hs on day 3. All patients will have iloperidone titrated to receive a dosage of at least 12 mg a day. Dosages can be titrated up to 24 mg a day based on tolerability and clinical indication. Dosage of iloperidone can be reduced to 6 mg a day if patients develop side effects necessitating a reduction in the dosage

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. Age 18 years and older
3. Patients on:

   * Li at a stable dose for 2 weeks or longer, and a serum level at screening of greater than or equal to 0.5 mEq/l OR
   * DIV dose for 2 weeks or longer, and a serum level at screening of greater than or equal to 45 ug/ml OR
   * LAM (dosage/day ≥100mg) at a stable dose for 2 weeks or longer OR
   * Any combination 3a, 3b, or 3c
4. Patients meeting DSM-IV TR diagnosis of bipolar disorder, I or II, as assessed using the MINI, (Sheehan et al., 1998) PLUS any ONE of criteria 5 or 6 or 7
5. Patients meeting DSM-IV TR diagnostic criteria for a mixed manic episode with Young Mania Rating Scale (YMRS) score>/=14 and Montgomery Asberg Depression Rating Scale (MADRS) score>/=14
6. Patients meeting the criteria for a manic/hypomanic episode for at least 2 days with the simultaneous presence of Young Mania Rating Scale (YMRS) score>/=14 PLUS Montgomery Asberg Depression Rating Scale (MADRS) score>/=14 ;
7. Patients meeting DSM-IV TR diagnostic criteria for a major depressive episode with the simultaneous presence of MADRS score>/=14 PLUS meeting the criteria for a manic/hypomanic episode for at least 2 days with the simultaneous presence of Young Mania Rating Scale (YMRS) score>/=14

Exclusion Criteria:

1. Patients with a current Axis I diagnosis of schizophrenia, schizophreniform disorder, schizotypal disorder, bipolar disorder with psychotic sub-type that requires hospitalization, drug induced mania or AIDS induced mania
2. Women with a positive pregnancy test or who are lactating
3. Women of child-bearing potential who are not practicing a clinically accepted method of contraception
4. Patients with general medical conditions that contraindicate psychoactive medications or uncontrolled medical disorder or central nervous system diseases.
5. Patients whose clinical status requires inpatient or day hospital treatment
6. History of severe side effects associated with therapeutic doses of Li, DIV, LAM
7. Alcohol or drug dependent at time of enrollment
8. Suicidal at time of enrollment.
9. Current or previous exposure to iloperidone
10. Patients taking medication that cause QTC prolongation
11. Patients with serious cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bowden, MD, Principal Investigator — UT Health Science Center San Antonio
Locations (1):
- UT Health Science Center San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred April 2013 to April 2015 from patients in the clinic or from responders to t.v. advertisements.
Pre-assignment Details: Subjects who met inclusion criteria at screening visit were started on study medication at visit 2.
Period: Overall Study
Arm/Group | Open Label Iloperidone
Started | 41
Completed | 16
Not Completed | 25

BASELINE CHARACTERISTICS:
Population: Subject meeting inclusion criteria
Arm/Group | Open Label Iloperidone
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Measure of Response by Change From Baseline to End of Study in BISS Depression and Mania Scale Scores
Description: The Bipolar Inventory of Symptoms Scale is a reliable and valid measure which assesses Depression and Mania symptoms of bipolar disorder. There are 42 items; each item is rated on a 0-4 scale. The BISS is a clinician-rated instrument. The Scale is rated as follows:
  0 Not at all
  1. Slight
  2. Mild
  3. Moderate
  4. Severe Each of the 42 items is rated separately, with a score, based on the most recent 7 day period.
  For Depression: Items 1-21 items of the assessment are summed up and multiplied by 4 to give a cumulative score out of 84. The higher the score, the more severe the depression.
  For Mania: Items 22-42 are summed up and multiplied by 4 to give a cumulative score out of 84. The higher the score, the more severe the mania. The mean is calculated from the change in score between baseline and week 20.
Time Frame: Baseline and 20 weeks
Population: Subjects who are currently treated with mood stabilizers (Lithium, Divalproex or Lamotrigine), with a diagnosis of Bipolar Disorder I or II.
Measure: Number; unit: percentage change in score on BISS scale
Groups:
- Mean Change in Depression for Study Completers: Measurement of mean change in depression for all subjects who entered study and completed 20 weeks
- Mean Change in Mania for Study Completers: Measurement of mean change in mania for all study participants who completed 20 weeks.
- Mean Change in Depression for All Study Participants: Mean change in depression for all study participants, including early terminators.
- Mean Change in Mania for All Study Participants: Mean change in mania for all study participants, including early terminators
Arm/Group | Mean Change in Depression for Study Completers | Mean Change in Mania for Study Completers | Mean Change in Depression for All Study Participants | Mean Change in Mania for All Study Participants
Number analyzed (Participants) | 16 | 16 | 41 | 41
percentage change in score on BISS scale | 35.7 | 61.8 | 25 | 48
Statistical Analysis 1: Comparison: Mean Change in Depression for Study Completers; BISS Outcomes: Mean changes in depression and mania for study completers were measured. The a priori hypothesis was a mean change of 50%; Test type: Superiority or Other; p < 0.0094, t-test, 2 sided — p value is not adjusted for multiple comparisons (see above). A priori threshold for significance was p<0.05; Mean Difference (Final Values) = -14.9, Standard Deviation 20.0
Statistical Analysis 2: Comparison: Mean Change in Mania for Study Completers; BISS Outcomes: Mean changes in mania for study completers were measured. The a priori hypothesis was a mean change of 50%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -15.4, Standard Deviation 10.1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Open Label Iloperidone
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 31/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Iloperidone (N=31)
dry mouth (Gastrointestinal disorders) | 12 (12)
dizzy/lightheaded (Nervous system disorders) | 8 (10)
Diarrhea/Loose stool (Gastrointestinal disorders) | 4 (4)
Heart palpitations (Cardiac disorders) | 9 (9)
Atrial fibrilation (Cardiac disorders) | 2 (2)
Flu symptoms/muscle weakness/fatigue (Immune system disorders) | 6 (8)
Anxiety (Psychiatric disorders) | 4 (4)
Nasal Congestion (Immune system disorders) | 5 (5)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Hypertension(high blood pressure) (Vascular disorders) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 8 (8)
weight gain (Metabolism and nutrition disorders) | 8 (8)
Decreased concertration (Psychiatric disorders) | 5 (5)
Increased Thirst (Endocrine disorders) | 11 (14)
Abdominal Bloating (Gastrointestinal disorders) | 2 (2)
Tremors (Musculoskeletal and connective tissue disorders) | 5 (5)
Edema of the legs (Blood and lymphatic system disorders) | 2 (2)
Drowsiness (General disorders) | 5 (5)
worsening of Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Blurry vision (Eye disorders) | 2 (2)
Migraine headache (Nervous system disorders) | 3 (3)
Dry Eyes (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No